CLINICAL TRIAL: NCT02685813
Title: Incidence of Pregnancies and Births With Spina Bifida in Denmark in 2008-2014
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aarhus University Hospital (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Charlotte Rosenkrantz Bodin, Medical and research year student, Aarhus University Hospital
Other Study IDs: SpinaBifida2016
Record Dates: First submitted 2016-02-11; First posted 2016-02-19 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Spina Bifida
Keywords: Ultra sound; birth defects
MeSH Terms: conditions — Spinal Dysraphism; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant women in Denmark: Pregnant women in Denmark participating in prenatal screening. This counts for approximately 50000 pregnancies/year and covers >95% of all pregnancies nationally.

SUMMARY:
Neural tube defects cover a group of severe embryo malformations such as anencephaly and spina bifida. The most severe forms of spina bifida causes numerous disabilities that demand lifelong treatment by a team consisting of primarily neurosurgeons, pediatricians, obstetricians, pediatric neurologists, pediatric urologists, gastroenterologists, psychologists and social workers. The disabilities involve morbidity such as decreased motor and sensory function caudal to the lesion, hydrocephalus, scoliosis, bladder and bowel incontinence as well as increased mortality.

In 2004, the Danish Health Authorities introduced new guidelines for fetal diagnostics. These represented a change of paradigm stating that all pregnant women should be offered a prenatal examination including an ultra sound scan in week 12-13 of gestation (including risk estimation of chromosomal diseases) as well as in week 19 of gestation (scanning primarily for malformations). The examination program was not elaborated to eradicate diseases but to support the reproductive autonomy of the pregnant women, including the possibility to seek for termination of the pregnancy in the case of severe disease in the fetus.

Severe spina bifida is one of the malformations that can be diagnosed with the ultra sound scan in week 19, and since the implementation of the new guidelines from the Danish Health Authority a study by this research group has shown decreased birth incidence at least in the Western part of Denmark.

It is still unknown what has caused this decrease as is the exact number of pregnancies and births complicated by spina bifida in the child; similarly it is unclear whether this decline is a regional or if it is only a Danish phenomenon.

By extraction of data from the Danish Fetal Database ("FØTOdatabasen") which includes information of all 60.000 pregnancies in Denmark annually, the purpose of this register study is to investigate the incidence of pregnancies complicated by prenatal diagnosis of spina bifida in Denmark from 2008 and on, as well as the pregnancy outcome in these cases (including termination of pregnancy). Furthermore results will be compared to results obtained by collaborative partners in Sweden and hopefully also in Saudi Arabia.

DETAILED DESCRIPTION:
Hypotheses:

The number of pregnancies in Denmark complicated by spina bifida in the child is constant, but the number of births in Denmark complicated by spina bifida in the child has declined, likely because the mother in most cases chooses to terminate the pregnancy in case of the diagnosis of severe spina bifida at the 19 week ultrasound scan.

Denmark is the only country in the world with a registered decline in the number of newborns with severe spina bifida.

Purpose:

1. Investigate the incidence of pregnancies complicated by prenatal diagnosis of spina bifida in Denmark from 2008 and on, as well as the pregnancy outcome in these cases (including termination of pregnancy).
2. In cooperation with international partners compare data from Denmark and Sweden (partner in Sweden: Eleonor Tiblad, MD, Ph.D, Center for Fetal Medicine, Karolinska University Hospital) and if possible also Saudi Arabia (partner in the Saudi Arabia collaboration: Marianne Juhler, MD, DMSc, Professor, Rigshospitalet, Denmark and Daniele Rigamonti, MD, professor, Chief of Staff, Department of Neurosurgery, John Hopkins University Hospital Aramco Health Care, Baltimore, USA)

Methods:

Regarding 1): Extraction of data from the Danish Fetal Database ("FØTOdatabasen") which includes information of all 60.000 pregnancies in Denmark annually.

Regarding 2): Data comparable to those collected in this study are expected to be delivered from collaborative partners in Sweden and Saudi Arabia. Comparison analysis of the data from our collaborative partners in Sweden and Saudi Arabia in order to discover differences in spina bifida pregnancy management on an international level.

Data from Saudi Arabia and Sweden:

The investigators will ask their partners in Sweden and Saudi Arabia to provide institutional, regional or national data comparable to those obtained in Denmark. Data from each pregnancy will then be compared on the following parameters:

* Prenatal diagnosis of spina bifida/MMC (ICD10: Q050-059)
* Pregnancy outcome: live birth, stillbirth, intrauterine death, spontaneous abortion, termination of pregnancy, fetal reduction in twin pregnancies
* Gestational age at outcome
* Epidemiological details of the cohort offered prenatal diagnostics (population based, institution based, population size
* Consultation guidelines and possibilities when spina bifida is diagnosed prenatally

The Danish Fetal Database:

FØTOdatabasen is a national fetal medicine database. The database includes information on maternal characteristics: age, parity, BMI, ethnicity, smoking status, Diabetes status (from 2014), and on the pregnancy: mode of conception, result of first trimester risk assessment for chromosomal anomalies, biometric data, ICD10-codes for any prenatally diagnosed malformation. FØTOdatabasen receives this information automatically on a daily basis from all birth departments' prenatal database (Astraia), and links data regarding each pregnancy with postnatal outcome from the Danish Cytogenetic Registry, the National Patient Registry and the National Birth Registry. FØTOdatabasen includes >95% of all pregnancies in Denmark with due date from 1. January 2008 and onwards. The data completeness is high, with missing data <1% for pregnancy outcome, <1% for smoking status, and <3% for mode of conception.

The database thereby provides a unique possibility to analyze population based data from approximately 55.0000 pregnancies annually with prenatal diagnosis and postnatal outcome. On an international level FØTOdatabasen thereby provides unique data to analyze pregnancies with spina bifida in a population and the pregnancy outcome, including live born children, intrauterine deaths and spontaneous as well as termination of pregnancy. Hereby it can be estimated how many incidences of spina bifida are isolated or associated with other malformations.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women, participating in prenatal screening

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: FØTOdatabasen is a national fetal medicine database, which includes information on maternal characteristics: age, parity, BMI, ethnicity, smoking status, diabetes status (from 2014), and on the pregnancy: mode of conception, result of first trimester risk assessment for chromosomal anomalies, biometric data, ICD10-codes for any prenatally diagnosed malformation. It links data regarding each pregnancy with postnatal outcome received from the Danish Cytogenetic Registry, the National Patient Registry and the National Birth Registry. FØTOdatabasen includes >95% of all pregnancies in Denmark with due date from 1. January 2008 and onwards. The data completeness is high, with missing data <1% for pregnancy outcome, <1% for smoking status, and <3% for mode of conception
Sampling Method: Non-Probability Sample
Enrollment: 350000 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-11 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
incidence of spina bifida | 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Olav B. Petersen, MD, ph.d, Study Director — Aarhus University Hospital; Mikkel M. Rasmussen, MD, ph.d, Study Chair — Aarhus University Hospital; Charlotte R. Bodin, Bsc.med, Principal Investigator — Aarhus University Hospital
Locations (1):
- Department of Gynecology and Obstetrics, Aarhus university Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Yes